CLINICAL TRIAL: NCT01912768
Title: Clinical Evaluation of the Safety and Efficacy of FID 120947A Compared to a Marketed Lens Care Solution
Brief Title: Safety and Efficacy Evaluation of a New Contact Lens Disinfecting Solution in Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: C-13-003
Record Dates: First submitted 2013-07-29; First posted 2013-07-31 (Estimated); Results first posted 2015-06-09 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-06

CONDITIONS: Myopia; Astigmatism; Hyperopia; Refractive Error
Keywords: contact lenses; contact lens solution; soft contact lenses
MeSH Terms: conditions — Myopia; Astigmatism; Hyperopia; Refractive Errors | interventions — Contact Lenses, Hydrophilic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- FID 120947A (Experimental): FID 120947A contact lens disinfecting solution used with soft contact lenses (study lenses) on a daily basis for 90 days
  Interventions: Device: FID 120947A contact lens disinfecting solution; Device: Soft contact lenses
- renu fresh (Active Comparator): Renu fresh multi-purpose solution used with soft contact lenses (study lenses) on a daily basis for 90 days
  Interventions: Device: renu fresh multi-purpose solution; Device: Soft contact lenses

INTERVENTIONS:
Device: FID 120947A contact lens disinfecting solution — Investigational 3% hydrogen peroxide solution intended for simultaneous cleaning, protein removal, disinfecting and storage of silicone hydrogel and soft contact lenses
  Other Names: Clear Care® Plus
  Arms: FID 120947A
Device: renu fresh multi-purpose solution — Commercially available solution indicated for cleaning, removing protein deposits, rinsing, chemical disinfection, and storage of soft contact lenses
  Arms: renu fresh
Device: Soft contact lenses — Commercially available soft contact lenses worn a minimum of 8 hours each day on a daily wear basis for the duration of the study (90 days). A fresh pair will be dispensed on Day 0, Day 30, and Day 60.

SUMMARY:
The purpose of this study is demonstrate substantial equivalence of an investigational contact lens disinfecting solution to a commercially available contact lens solution in silicone hydrogel and soft contact lens wearers.

DETAILED DESCRIPTION:
Subjects with normal eyes (other than correction for refractive error) successfully wearing soft contact lenses were randomized 2:1 to receive either the investigational or commercial contact lens solution for daily use throughout the study (90 days).

ELIGIBILITY:
Inclusion Criteria:

* Normal eyes (other than correction for visual acuity);
* Successful history of silicone hydrogel or soft contact lens wear in both eyes in one of the following brands: Soflens® 38, Proclear DW, Frequency 55, Acuvue® Oasys™, Air Optix Aqua, O2 OPTIX, Air Optix for Astigmatism, Air Optix Aqua Multifocal, Biofinity®, PureVision®, PureVision®2;
* Best spectacle corrected distance visual acuity greater than or equal to 20/25 in each eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any ocular or systemic medical condition that may, in the opinion of the investigator, preclude safe administration of the investigational products or affect the results of this study;
* Need to wear contact lenses on an extended wear basis (ie, overnight) during the study;
* Use of a daily cleaner and/or an enzyme cleaner to care for lenses at least 7 days prior to Visit 1;
* History of intolerance or hypersensitivity to any component of the investigational products;
* Use of all over-the-counter (OTC) or prescribed topical ocular medications within 7 days prior to Visit 1;
* Moderate, severe, abnormal, or other ocular findings;
* Current or history of ocular infection, severe inflammation, or disease within 6 months prior to Visit 1;
* Any systemic disease at Visit 1 (including allergies, respiratory infections or colds) that may affect the eye or be exacerbated by use of contact lenses or contact lens solutions;
* Use of systemic medications that may contribute to adverse ocular effects unless on a stable dosing regimen;
* Ocular surgery within the last 12 months;
* Other protocol-defined exclusion criteria may apply.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2013-12; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Monica Studzinski, Lead CSM, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 17 study centers located in the US.
Pre-assignment Details: Of the 362 enrolled, 10 subjects were exited as screen failures prior to randomization. This reporting group includes all randomized subjects (352).
Groups:
- FID 120947A: Contact lens disinfecting solution used with soft contact lenses (study lenses) on a daily basis for 90 days
- Renu Fresh: Multi-purpose solution used with soft contact lenses (study lenses) on a daily basis for 90 days
Period: Overall Study
Arm/Group | FID 120947A | Renu Fresh
Started | 239 | 113
Completed | 229 | 109
Not Completed | 10 | 4
Not completed — Adverse Event | 2 | 0
Not completed — Lost to Follow-up | 2 | 1
Not completed — Withdrawal by Subject | 5 | 3
Not completed — Randomized in error | 1 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | FID 120947A | Renu Fresh | Total
Number analyzed (Participants) | 239 | 113 | 352
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (11.7) | 35.3 (10.9) | 34.8 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 92 | 266
  Male | 65 | 21 | 86

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Visibly Clean Lenses
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. A lens was considered visibly clean if it had nondetectable films or deposits. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all randomized subjects. Here, "n" is the total number of subjects with data in each treatment group, respectively, by visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, n=236, 113 | 44.5 | 39.8
  Day 30, n=234, 112 | 35.0 | 31.3
  Day 60, n=232, 110 | 40.5 | 32.7
  Day 90, n=229, 109 | 41.9 | 33.0

2. Primary Outcome: Percentage of Subjects With Crystalline Deposits by Type
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered: Type II = films or deposits visible only under special conditions, such as special illumination using an eyepiece of 7-10 times magnification, Type III = films or deposits readily visible on a dry lens under room lighting, with unaided eye, and Type IV = films or deposits obvious under room lighting, with unaided eye, when the lens is wet or dry. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all randomized subjects. Here, "n" is the total number of subjects with crystalline deposits in each treatment group, respectively, by visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, Type II, n=55,32 | 63.6 | 65.6
  Day 7, Type III, n=55,32 | 25.5 | 25.0
  Day 7, Type IV, n=55,32 | 10.9 | 9.4
  Day 30, Type II, n=74, 37 | 70.3 | 59.5
  Day 30, Type III, n=74, 37 | 10.8 | 16.2
  Day 30, Type IV, n=74, 37 | 18.9 | 24.3
  Day 60, Type II, n=73, 36 | 63.0 | 41.7
  Day 60, Type III, n=73, 36 | 13.7 | 25.0
  Day 60, Type IV, n=73, 36 | 23.3 | 33.3
  Day 90, Type II, n=69, 42 | 60.9 | 59.5
  Day 90, Type III, n=69, 42 | 18.8 | 19.0
  Day 90, Type IV, n=69, 42 | 20.3 | 21.4

3. Primary Outcome: Percentage of Subjects With Film Deposits by Type
Description: as for outcome 2
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: This analysis population includes all randomized subjects. Here, "n" is the total number of subjects with film deposits in each treatment group, respectively, by visit.
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, Type II, n=114, 56 | 57.0 | 58.9
  Day 7, Type III, n=114, 56 | 16.7 | 19.6
  Day 7, Type IV, n=114, 56 | 26.3 | 21.4
  Day 30, Type II, n=125, 66 | 62.4 | 62.1
  Day 30, Type III, n=125, 66 | 14.4 | 13.6
  Day 30, Type IV, n=125, 66 | 23.2 | 24.2
  Day 60, Type II, n=114, 63 | 63.2 | 55.6
  Day 60, Type III, n=114, 63 | 8.8 | 7.9
  Day 60, Type IV, n=114, 63 | 28.1 | 36.5
  Day 90, Type II, n=114, 59 | 64.9 | 50.8
  Day 90, Type III, n=114, 59 | 10.5 | 13.6
  Day 90, Type IV, n=114, 59 | 24.6 | 35.6

4. Primary Outcome: Average Residual Lens Lysozyme
Description: Worn study lenses were removed and analyzed by high performance liquid chromatography (HPLC) for residual lens lysozyme (protein). Values reported as lower than the limit of quantitation or none detected were imputed as 0.5 μg or 0 μg, respectively. A lower value indicates less lysozyme deposition. One eye (study eye) contributed to the analysis.
Time Frame: Day 30/Early Exit
Population: This analysis population includes all subjects with data at visit.
Measure: Mean (Standard Deviation); unit: micrograms per lens
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 233 | 112
micrograms per lens | 70.2 (192.1) | 114.5 (295.5)

5. Primary Outcome: Percentage of Subjects With Change From Baseline in Contact Lens-Corrected Distance Visual Acuity (CLCDVA) by Line Change
Description: Distance VA was assessed for each eye individually while reading a chart distant to the participant in dimmed room illumination. VA was measured using a Snellen chart, with 20/20 Snellen acuity considered normal distance-eyesight. A line increase indicates an improvement in VA. One eye (study eye) contributed to the analysis.
Time Frame: Baseline (Day 0), Day 7, Day 30, Day 60, Day 90
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, 2 Line Increase from Baseline, n=236, 112 | 0.0 | 0.0
  Day 7, 1 Line Increase from Baseline, n=236, 112 | 0.4 | 0.9
  Day 7, No Change from Baseline, n=236, 112 | 97.0 | 99.1
  Day 7, 1 Line Decrease from Baseline, n=236, 112 | 2.5 | 0.0
  Day 7, 2 Line Decrease, n=236, 112 | 0.0 | 0.0
  Day 30, 2 Line Increase from Baseline, n=234, 112 | 0.0 | 0.0
  Day 30, 1 Line Increase from Baseline, n=234, 112 | 2.1 | 0.0
  Day 30, No Change from Baseline, n=234, 112 | 95.7 | 99.1
  Day 30, 1 Line Decrease from Baseline, n=234, 112 | 2.1 | 0.9
  Day 30, 2 Line Decrease from Baseline, n=234, 112 | 0.0 | 0.0
  Day 60, 2 Line Increase from Baseline, n=232, 110 | 0.0 | 0.0
  Day 60, 1 Line Increase from Baseline, n=232, 110 | 1.7 | 0.0
  Day 60, No Change from Baseline, n=232, 110 | 95.7 | 98.2
  Day 60, 1 Line Decrease from Baseline, n=232, 110 | 2.6 | 1.8
  Day 60, 2 Line Decrease from Baseline, n=232, 110 | 0.0 | 0.0
  Day 90, 2 Line Increase from Baseline, n=229, 109 | 0.0 | 0.0
  Day 90, 1 Line Increase from Baseline, n=229, 109 | 2.2 | 0.0
  Day 90, No Change from Baseline, n=229, 109 | 94.3 | 98.2
  Day 90, 1 Line Decrease from Baseline, n=229, 109 | 3.1 | 1.8
  Day 90, 2 Line Decrease from Baseline, n=229, 109 | 0.4 | 0.0

6. Primary Outcome: Average Lens Wear Time
Description: Subject recorded a response to the question, "Averaging over the last 3 days, how many hours per day did you wear your contact lenses?" Lens wear time was measured in hours.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
Hours
  Day 7, n=236, 113 | 12.9 (2.6) | 12.6 (2.6)
  Day 30, n=234, 112 | 12.9 (2.7) | 12.6 (2.6)
  Day 60, n=232, 110 | 13.0 (2.6) | 12.6 (2.6)
  Day 90, n=229, 109 | 13.1 (2.7) | 12.9 (2.7)

7. Primary Outcome: Number of Unscheduled Lens Replacements by Reason
Description: A fresh pair of lenses was dispensed on Day 0, Day 30, and Day 60. Lenses replaced at other times were considered unscheduled. The counts in the table represent the total number of unscheduled lenses replaced by reason for any eye, any subject.
Time Frame: Up to Day 90
Population: This analysis population includes all randomized subjects.
Measure: Number; unit: lenses
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
lenses
  Discomfort | 3 | 0
  Lost | 4 | 0
  Lens torn on eye | 2 | 0
  Lens torn while handling | 5 | 5
  Other | 9 | 7

8. Primary Outcome: Likert Item - "When I Use This Solution, my Lenses Are Comfortable All Day."
Description: Lens comfort was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, Strongly Agree, n=236, 113 | 30.1 | 36.3
  Day 7, Agree, n=236, 113 | 55.1 | 50.4
  Day 7, Undecided, n=236, 113 | 5.1 | 3.5
  Day 7, Disagree, n=236, 113 | 8.9 | 7.1
  Day 7, Strongly Disagree, n=236, 113 | 0.8 | 2.7
  Day 30, Strongly Agree, n=234, 112 | 29.9 | 24.1
  Day 30, Agree, n=234, 112 | 50.9 | 51.8
  Day 30, Undecided, n=234, 112 | 5.1 | 6.3
  Day 30, Disagree, n=234, 112 | 12.0 | 16.1
  Day 30, Strongly Disagree, n=234, 112 | 2.1 | 1.8
  Day 60, Strongly Agree, n=232, 110 | 24.6 | 21.8
  Day 60, Agree, n=232, 110 | 54.3 | 51.8
  Day 60, Undecided, n=232, 110 | 6.5 | 5.5
  Day 60, Disagree, n=232, 110 | 13.8 | 14.5
  Day 60, Strongly Disagree, n=232, 110 | 0.9 | 6.4
  Day 90, Strongly Agree, n=229, 109 | 28.8 | 23.9
  Day 90, Agree, n=229, 109 | 54.6 | 59.6
  Day 90, Undecided, n=229, 109 | 4.8 | 5.5
  Day 90, Disagree, n=229, 109 | 10.5 | 9.2
  Day 90, Strongly Disagree, n=229, 109 | 1.3 | 1.8

9. Primary Outcome: Likert Item - "When I Use This Solution, at the End of the Lens Wearing Day my Vision is Clear."
Description: Clear vision was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, Strongly Agree, n=236, 113 | 30.5 | 29.2
  Day 7, Agree, n=236, 113 | 57.2 | 59.3
  Day 7, Undecided, n=236, 113 | 6.4 | 6.2
  Day 7, Disagree, n=236, 113 | 5.5 | 4.4
  Day 7, Strongly Disagree, n=236, 113 | 0.4 | 0.9
  Day 30, Strongly Agree, n=234, 112 | 27.4 | 20.5
  Day 30, Agree, n=234, 112 | 53.8 | 59.8
  Day 30, Undecided, n=234, 112 | 5.1 | 7.1
  Day 30, Disagree, n=234, 112 | 12.4 | 9.8
  Day 30, Strongly Disagree, n=234, 112 | 1.3 | 2.7
  Day 60, Strongly Agree, n=232, 110 | 20.3 | 17.3
  Day 60, Agree, n=232, 110 | 62.1 | 61.8
  Day 60, Undecided, n=232, 110 | 5.2 | 6.4
  Day 60, Disagree, n=232, 110 | 12.1 | 11.8
  Day 60, Strongly Disagree, n=232, 110 | 0.4 | 2.7
  Day 90, Strongly Agree, n=229, 109 | 24.5 | 17.4
  Day 90, Agree, n=229, 109 | 59.4 | 63.3
  Day 90, Undecided, n=229, 109 | 6.6 | 7.3
  Day 90, Disagree, n=229, 109 | 9.2 | 8.3
  Day 90, Strongly Disagree, n=229, 109 | 0.4 | 3.7

10. Primary Outcome: Likert Item - "When I Use This Solution, I Like the Way This Product Feels During Handling."
Description: Product handling was assessed by the subject as a single response on a 5-point Likert scale (Strongly Agree, Agree, Undecided, Disagree, Strongly Disagree) to best describe their lens wearing experience over the last 3 days. Responses were summarized by agreement category and presented as percentage of subjects.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of subjects
  Day 7, Strongly Agree, n=236, 113 | 31.4 | 38.1
  Day 7, Agree, n=236, 113 | 52.1 | 47.8
  Day 7, Undecided, n=236, 113 | 10.2 | 6.2
  Day 7, Disagree, n=236, 113 | 5.9 | 4.4
  Day 7, Strongly Disagree, n=236, 113 | 0.4 | 3.5
  Day 30, Strongly Agree, n=234, 112 | 27.8 | 25.0
  Day 30, Agree, n=234, 112 | 59.0 | 59.8
  Day 30, Undecided, n=234, 112 | 9.0 | 6.3
  Day 30, Disagree, n=234, 112 | 3.0 | 8.0
  Day 30, Strongly Disagree, n=234, 112 | 1.3 | 0.9
  Day 60, Strongly Agree, n=232, 110 | 25.0 | 28.2
  Day 60, Agree, n=232, 110 | 62.5 | 51.8
  Day 60, Undecided, n=232, 110 | 6.5 | 10.0
  Day 60, Disagree, n=232, 110 | 4.7 | 8.2
  Day 60, Strongly Disagree, n=232, 110 | 1.3 | 1.8
  Day 90, Strongly Agree, n=229, 109 | 28.4 | 28.4
  Day 90, Agree, n=229, 109 | 60.7 | 56.0
  Day 90, Undecided, n=229, 109 | 4.8 | 7.3
  Day 90, Disagree, n=229, 109 | 4.8 | 6.4
  Day 90, Strongly Disagree, n=229, 109 | 1.3 | 1.8

11. Primary Outcome: Crystalline Deposit Area Covered
Description: Worn study lenses were removed and evaluated for deposits. Deposits found on the lenses were defined using a 3-part classification system consisting of general visibility, the specific appearance and area covered. Values were reported as a percentage of lens area covered. One eye (study eye) contributed to the analysis.
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of lens area
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of lens area
  Day 7, n=55, 32 | 12.5 (12.2) | 17.8 (18.5)
  Day 30, n=74, 37 | 12.1 (9.8) | 14.0 (16.8)
  Day 60, n=73, 36 | 13.0 (10.2) | 13.3 (10.2)
  Day 90, n=69, 42 | 12.2 (10.9) | 14.0 (15.1)

12. Primary Outcome: Film Deposit Area Covered
Description: as for outcome 11
Time Frame: Day 7, Day 30, Day 60, Day 90
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: percentage of lens area
Arm/Group | FID 120947A | Renu Fresh
Number analyzed (Participants) | 239 | 113
percentage of lens area
  Day 7, n=114, 56 | 18.7 (12.2) | 16.7 (12.1)
  Day 30, n=125, 66 | 18.9 (14.3) | 20.5 (14.4)
  Day 60, n=114, 63 | 21.0 (16.1) | 23.4 (15.3)
  Day 90, n=114, 59 | 17.3 (12.8) | 20.9 (14.6)

ADVERSE EVENTS:
Time Frame: An Adverse Event (AE) was any untoward medical occurrence, unintended disease or injury, or untoward clinical signs in subjects, whether or not related to the investigational medical device. AEs are reported as pre-treatment and treatment-emergent.
Description: AEs were collected for the duration of the study (Dec 2013-May 2014). AEs were obtained as solicited and volunteered comments from subjects and as observations by the Investigator as outlined in the protocol. One subject was randomized but never received investigational product and was excluded from the safety dataset.
Groups:
- Pre-treatment: All subjects who consented to participate in the study prior to exposure to investigational product
- FID 120947A: All subjects who were exposed to FID 120947A
- Renu Fresh: All subjects who were exposed to renu fresh
Arm/Group | Pre-treatment | FID 120947A | Renu Fresh
Serious Adverse Events (participants affected / at risk) | 0/362 | 1/238 | 0/113
Other Adverse Events (participants affected / at risk) | 0/362 | 0/238 | 0/113
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-treatment (N=362) | FID 120947A (N=238) | Renu Fresh (N=113)
ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.